CLINICAL TRIAL: NCT05623241
Title: PERSPECTIVE MONOCENTRIC STUDY: USE OF LIQUID BIOPSY AND DIAGNOSTIC IMAGING IN THE SEARCH FOR CIRCULATING TUMOR DNA IN PATIENTS WITH BREAST CANCER
Brief Title: MONOCENTRIC PERSPECTIVE STUDY: USE OF LIQUID BIOPSY WITH DIAGNOSTIC IMAGING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gianluca Gatta, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 0023041/i
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Liquid Biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy — Venous blood sampling for liquid biopsy in breast cancer patients after segmentation of the lesion on mammography

SUMMARY:
Evaluation of the diagnostic accuracy of Mammography in the morpho-structural analysis of mammographic images in breast cancer-diagnosed patients or patients in follow-up for breast cancer by extracting a number of features describing the texture and morphology of the lesions reported in the form of a structured report explicitly developed for the study. Correlation of the data obtained from evaluating the primary endpoint with the genetic/molecular analysis on liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

* full information on the study and signature of the informed consent
* biopsy-proven breast cancer or previous surgery for breast cancer
* willingness of the patient to undergo liquid biopsy

Exclusion Criteria:

* state of pregnancy or breastfeeding
* patients operated on for benign or inflammatory diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are enrolled in mammography screening
Study Population: The liquid biopsy will be performed on all patients who undergo a mammography examination in which a malignant focal aspect has been found and who agree to participate in the study. All patients enrolled in the study will be subjected to a peripheral venous blood sample. The ctDNA will be extracted for molecular analysis and will be performed with NGS (Next Generation Sequencing) technology.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Radiomic of breast cancers and liquid biopsy | 36 months
  Detect possible relationships between breast cancers radiomic feature and genetic mutations on liquid biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- University "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided